CLINICAL TRIAL: NCT03254199
Title: A Randomized, Double-Blind, Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of FLX-787-ODT for Treatment of Muscle Cramps in Adult Subjects With Charcot-Marie-Tooth Disease
Brief Title: A Study to Assess the Safety and Effectiveness of FLX-787 in Subjects With Charcot-Marie-Tooth Disease Experiencing Muscle Cramps.
Acronym: COMMIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor
Sponsor: Flex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLX-787-204
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Charcot-Marie-Tooth Disease
Keywords: Charcot-Marie-Tooth; CMT; Muscle Cramps; Muscle Cramping; FLX-787; Hereditary Sensory and Motor Neuropathy; Neurogenetic disorder; Nervous System Malformations; Nervous System Diseases; Neurodegenerative Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Muscle Cramp; Spasm; Hereditary Sensory and Motor Neuropathy; Nervous System Malformations; Nervous System Diseases; Neurodegenerative Diseases; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: FLX-787-ODT (orally disintegrating tablet)
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo ODT

INTERVENTIONS:
Drug: FLX-787-ODT (orally disintegrating tablet) — FLX-787-ODT taken three times daily for 28 days
  Arms: Experimental
Drug: Placebo ODT — Placebo ODT taken three times daily for 28 days
  Arms: Placebo Comparator

SUMMARY:
The COMMIT Study will assess the safety and effectiveness of FLX-787 in men and women with Charcot-Marie-Tooth disease (CMT) experiencing muscle cramps. Participants will be asked to take two study products during the course of the study. One of these study products will be a placebo.

Approximately 120 participants in 20 study centers across the United States are expected to take part. Participants will be in the study for approximately 3 months and visit the study clinic 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptoms of CMT since at least 6 months prior to Screening, and confirmed diagnosis of CMT as defined by:

  1. Genetic confirmation of a mutation known to cause CMT, or
  2. Clinical and electrophysiological evidence of CMT and a genetic confirmation in a family member. Clinical features include length dependent sensory and motor loss, with sensorimotor axonal or demyelinating changes on a nerve conduction study.
* Weekly muscle cramping (defined as: a sustained muscle contraction that's most often painful and lasts seconds to minutes)

Exclusion Criteria:

* Presence of major gastrointestinal disorders, such as inflammatory bowel disease, diverticulitis, active peptic ulcer disease, or significant gastroesophageal reflux disease (i.e., not well-controlled on antacids or proton pump inhibitors), or oral or esophageal lesions/ulcers
* Presence of significant swallowing problems
* Unable or unwilling to discontinue medications for cramps and/or opiates
* Inability to tolerate a spicy sensation in the mouth or stomach
* Actively using illicit drugs or history of chronic substance abuse within the past year prior to screening, including abuse of alcohol
* Intention to change the current level of tobacco use or use of nicotine-containing products (i.e., new smokers or those actively trying to quit may not enrolled)
* Participated in a clinical study (except natural history studies without administration of an investigational product) within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Cramp frequency | 28 days
  Cramp frequency measured over the 28-day treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Johnson, MD, Principal Investigator — University of Utah
Locations (20):
- United States (20):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brighman and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - The University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Saint Luke's Rehabilitation Institute, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided